CLINICAL TRIAL: NCT01997320
Title: Effect of Strength Training and Protein Supplementation on the Muscle Function in Very Old Nursinghome Residents
Brief Title: Effect of Strength Training and Protein Supplementation on Muscles in the Very-old
Acronym: 83+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Leidersdorff Bechshøft, M.D., Ph.d. student, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-4-2013-068
Record Dates: First submitted 2013-11-11; First posted 2013-11-28 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Ageing
Keywords: Sarcopenia; Frailty; Strength; Protein supplementation; Ageing
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heavy resistance exercise and nutrition (Experimental): Heavy resistance exercise of the lower extremities three times weekly for 12 weeks combined with nutrient supplementation twice daily each containing 20g of milk protein.
  Interventions: Other: Heavy resistance exercise and nutrition
- Nutrition supplement (Active Comparator): Nutrient supplementation twice daily for 12 weeks. Each supplement contains 20g of milk protein.
  Interventions: Other: Nutrition supplement

INTERVENTIONS:
Other: Heavy resistance exercise and nutrition — Heavy resistance exercise of the lower extremities three times weekly for 12 weeks.
  Arms: Heavy resistance exercise and nutrition
Other: Nutrition supplement — Two daily administrations of nutrient supplementation, each containing 20g of milk protein.
  Arms: Nutrition supplement

SUMMARY:
Three months intervention study, investigating the effect of nutrient supplementation (including 20g of milk protein) twice daily with or without additional heavy resistance exercise three times weekly on muscle size, structure and function in 30 subjects at least 83 years of age.

Primary hypothesis is that the group conducting exercise improves muscle size, structure and function.

DETAILED DESCRIPTION:
A total of 30 subjects at least 83 years of age are recruited using advertisements in newspapers, magazines, public places and further personal contact. After information and written ethical consent (in accordance with the Declaration of Helsinki II) health status is evaluated by a medical doctor including blood screening, screening for dementia and routine objective evaluation. If there is no reason to exclude subjects (see exclusion criteria), they are whole-body DXA-scanned (Dual X-ray Absorptiometry) and MR-scanned (Magnetic resonance imaging)(dominant knee and femur) and functional measures (30s chair-stand, 10m and 8m gait speed, DEMMI-test) and strength measures (isometric and isokinetic leg power, power rig, grip strength) and tendon stiffness are measured. At least 4 days after this the first muscle biopsy in the dominant m. vastus lateralis is taken. Hereafter subjects are randomized to one of two groups:

Group one (n=15) is the exercise and nutrition group (HRT). Subjects in this group are to conduct supervised center-based heavy resistance exercise of the lower extremities three times weekly for 12 weeks. As for group two, this group receives nutritional supplementation twice daily throughout the 12 weeks period. Supplementation contains 20g of milk protein and some carbohydrate and lipids.

Group two (n=15) is the nutrition group (PRO). Subjects in this group only receives nutritional supplementation as described above.

After 12 weeks of intervention the same strength- and functional measures are made, DXA- and MR-scans and a second biopsy is made along with tendon stiffness measurement.

Data is collected and analyzed by staff blinded to randomization. Personal data is locked up, and only anonymized data is analyzed. Differences in both primary (m. quadriceps femoris cross sectional area) and secondary outcomes (functional measures, strength measures, muscle cell- and fiber type count, mRNA expression, muscle collagen content and distribution) are evaluated using two-way anova with repeated measures and, if allowed, post-hoc tests. Analysis will be made as intention-to-treat.

Power:

With an expected 10% increase in quadriceps CSA (cross-sectional area) (from 4500 square mm at baseline) with a SD of 600 square mm, power is 82% with alfa 0.05 with inclusion of 15 subjects in each group.

In case of systematic health-issues in response to the intervention, the trial will end immediately.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 83 years

Exclusion Criteria:

* Acute severe medical or surgical illnesses.
* Unstable chronic diseases, eg. renal failure, uncontrolled cardiac arrythmias, severe COPD (Chronic Obstructive Pulmonary Disease), diabetes mellitus.
* Bilateral knee alloplastics
* Metal devices compromising MR-scanning.
* Medicine: Anticoagulants (K-vitamin antagonists, heparins, ADP-receptor blockers, direct thrombin inhibitors, factor Xa inhibitors), systemic steroid treatment.
* Dementia
* Regular heavy load resistance exercise more than 20 min/week.

Min Age: 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps muscle cross sectional area from baseline to 3 months | 0 and 3 months
  Assessed by MRI scanning of dominant thigh. 8 slices, each of 1cm thickness, separated by 5cm.

SECONDARY OUTCOMES:
Change in isometric muscle strength from baseline to 3 months | 0 and 3 months
  Unilateral measurement of isometric strength in m. quadriceps femoris using KinCom.
Change in isokinetic muscle strength from baseline to 3 months | 0 and 3 months
  Unilateral isokinetic muscle strength at 60 degrees/s of m. quadriceps femoris.
Change in leg power from baseline to 3 months | 0 and 3 months
  Using a Powerrig, unilateral leg extension power is determined.

OTHER OUTCOMES:
Change in gait speed from baseline to 3 months | 0 and 3 months
  Gait speed averaged over 10m including acceleration. Gait speed averaged over 8m excluding acceleration.
Change in DEMMI from baseline to 3 months | 0 and 3 months
  DeMorton Mobility Index
Change in 30s chair-stand from baseline to 3 months | 0 and 3 months
  30s chair-stand
Change in Short Form-36 questionnaire from baseline to 3 months | 0 and 3 months
Change in patella tendon stiffness from baseline to 3 months | 0 and 3 months
  Stress-deformation of dominant patella tendon using ultrasound.
Change in muscle biopsy from baseline to 3 months | 0 and 3 months
  Measurements of fiber types, size, capillary density, satellite cell count, mRNA-targets, western blotting, muscular collagen content and distribution.
Change in standard health parameters from baseline to 3 months | 0 and 3 months
  Blood pressure, plasma lipids, HbA1c, anthropometry

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, MD, Proff., Study Chair — Head of department
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispbebjerg Hospital, Copenhagen NV, Denmark, Denmark